CLINICAL TRIAL: NCT06791577
Title: Bridging the Healing Gap: A Single-Blind Clinical Trial Assessing the Efficacy of Carboxy-gel in Reducing Bruising and Pain Post-Liposuction
Acronym: CO2L001
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Total Definer Research Group (Other)
Responsible Party: Principal Investigator, Alfredo Hoyos, Plastic Surgeon, Total Definer Research Group
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Carboxy-gel (CO2 Lift)
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Liposuction; Bruising; Inflammation; Pain, Postoperative; Ecchymosis; Hematoma
Keywords: Carboxytherapy; CO2 Lift; Body contouring; Liposuction; Liposculpture; High Definition Liposculpture; Patient outcomes
MeSH Terms: conditions — Contusions; Inflammation; Pain, Postoperative; Ecchymosis; Hematoma

STUDY DESIGN:
Intervention Model Description: Each patient serves as their own control, with one area receiving the intervention (CO2 Lift) and the contralateral area receiving placebo (Vaseline)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 Lift group (Experimental): * Application of CO2 lift to one arm, and/or one glute, and/or one half of the lower abdomen.
  * Apply immediately after surgery and 12 hours later. Then one time per day for 3-5 days for patients with low risk for flap/skin ischemia/suffering.
  Interventions: Drug: Carboxytherapy
- Control group (Placebo Comparator): * Application of Vaseline to the contralateral area in which CO2 lift was applied, using the same timing protocol as per CO2 lift
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Carboxytherapy — Application of the intervention (CO2 Lift) in the area according to the protocol schedule
  Arms: CO2 Lift group
Other: Placebo — Application of the placebo (Vaseline) in the area according to the protocol schedule
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate if CO2 Lift reduces bruising and pain after Liposuction. The study also aims to explore changes in patient satisfaction. The main questions this study seeks to answer are:

* Does CO2 lift reduce the extent of bruising at 7 days post-surgery?
* How does CO2 lift impact patient-reported pain and satisfaction?

In this study, researchers will compare CO2 lift to a placebo (Vaseline) to see if the intervention has a positive effect.

The study procedures include:

* Baseline data collection of sociodemographic variables. Data collection of surgical variables, adverse events, pain scores, and satisfaction scores.
* During the liposuction procedure the patient will receive CO2 Lift application to one arm, and/or one glute, and/or one half of the lower abdomen, and placebo (Vaseline) to the contralateral part.
* Apply CO2 lift and Vaseline immediately after surgery, 12 hours later, and then once a day for 3 to 5 days depending of the risk of the flap/skin.
* Postoperative follow-up with photos of treated areas at 24 hours, 3 days, and 7 days, with bruising quantified using Image J software.

DETAILED DESCRIPTION:
Study Design: Randomized, controlled, single-blind trial

* Allocation: Randomized (one area with CO2 lift treatment, one area with Vaseline control)
* Intervention Model: Comparative contralateral randomized clinical trial (each participant serves as their own control, with CO2 lift applied to one area and Vaseline to the contralateral area).
* Masking: Single-blind (Participants are blinded to the treatment allocation).

Study Locations:

* Dhara Clinic, Bogota, Colombia
* Private Practice, Sao Paulo, Brazil
* Private Practice, Mexico City, Mexico

Data Collection:

* Photographic analysis with ImageJ, from photo records from days 1, 3, 7 post procedure, to calculate the percentage of the area with ecchymosis.
* Pain Assessment: Visual Analogue Scale (VAS) scores recorded at the same time points.
* Satisfaction Scores: Global Aesthetic Improvement Scale (GAIS) evaluated at least 3 months postoperatively.

Ethical Considerations:

* Informed Consent: Participants will be provided comprehensive information about study procedures, risks, and benefits, and written consent will be obtained.
* IRB Approval: The study will adhere to the Declaration of Helsinki principles and will be approved by an Institutional Review Board (IRB).
* Data Confidentiality: All participant data will be anonymized and securely stored.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing body contouring procedures (liposuction or liposculpture), either individually or combined with a maximum of two other major aesthetic procedures involving face, breast, or dermo-lipectomy.
* healthy patients without underlying comorbidities (classified as ASA≤II)

Exclusion Criteria:

* Pregnant patients
* Known allergy to CO2 Lift or Vaseline
* History of keloid formation or significant dermatological conditions.
* Coagulopathy or current use of anticoagulant therapy.
* Skin disorders related to collagen disease.
* BMI ≥ 32 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Ecchymosis of the area - 7 days post procedure | 7 days
  Reduction of ecchymosis in each area, measured using Photomicrographic analysis with ImageJ Software. The unit of measurement will me in cm^2 of the affected area (bruised) normalized to the total area of the area (in cm^2).

SECONDARY OUTCOMES:
Ecchymosis of the area - 24 hours post procedure | 24 hours
  Reduction of ecchymosis in each area, measured using Photomicrographic analysis with ImageJ Software. The unit of measurement will me in cm^2 of the affected area (bruised) normalized to the total area of the area (in cm^2).
Ecchymosis of the area - 3 days post procedure | 3 days
  Reduction of ecchymosis in each area, measured using Photomicrographic analysis with ImageJ Software. The unit of measurement will me in cm^2 of the affected area (bruised) normalized to the total area of the area (in cm^2).
Pain Score | 7 days
  Patient-reported pain measured using Pain Visual Analogue Scale (VAS), measured at 24 hours, 3 days, and 7 days post-procedure. In the VAS pain scores, 0 represents no pain, while 10 represents the worst possible pain experienced.
Patient Satisfaction Scores | 6 months
  Patient reported satisfaction scores measured using Global Aesthetic Improvement Scale (GAIS).
  The GAIS is a standardized scale used primarily in cosmetic and dermatological treatments to assess the overall aesthetic improvement of a patient after a procedure. It consist of three questions: * how do you feel about your appearance after surgery? Possible answers: Very much improved, much improved, slightly improved, no change. * Are you satisfied with the surgery? Very satisfied, satisfied, not satisfied. * Would you recommend the surgical procedure? Possible answers: Yes, perhaps, no.

CONTACTS AND LOCATIONS:
Locations (3):
- Private Practice, São Paulo, Brazil
- Dhara clinic, Bogotá, DC, Colombia
- Private Practice, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Depending upon reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately after publication.
Access Criteria: Request to the main author

REFERENCES:
- [Background] Oliveira SMD, Rocha LB, da Cunha MTR, Cintra MMM, Pinheiro NM, Mendonca AC. Effects of carboxytherapy on skin laxity. J Cosmet Dermatol. 2020 Nov;19(11):3007-3013. doi: 10.1111/jocd.13337. Epub 2020 Feb 24. PMID 32091181
- [Background] Delgado-Miguel C, Miguel-Ferrero M. Preliminary results of the use of carboxytherapy in the treatment of pathologic scars: A minimally invasive alternative. J Pediatr Surg. 2023 Apr;58(4):679-683. doi: 10.1016/j.jpedsurg.2022.12.008. Epub 2022 Dec 22. PMID 36641310
- [Background] Waked K, Kierdaj M, Aslani A. The Use of Carboxytherapy for the Treatment of Deep Partial-Thickness Skin Burns After Circumferential and High-Definition Liposuction: Promising Clinical Results in 5 Consecutive Cases. Aesthetic Surg J Open Forum. 2023;5:ojad096. doi:10.1093/asjof/ojad096